CLINICAL TRIAL: NCT00003250
Title: Phase I Evaluation of Fenretinide (NSC# 374551)
Brief Title: Fenretinide in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066130; U01CA062487 (NIH); P30CA022453 (NIH); WSU-C-1605; NCI-T97-0098
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of fenretinide in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and toxicity of oral fenretinide in patients with solid malignant tumors. II. Determine the pharmacokinetics of fenretinide and its metabolites. III. Determine the preliminary antitumor activity of fenretinide in this patient population. IV. Determine the recommended phase II starting dose of fenretinide. V. Determine whether fenretinide induces apoptosis in clinical specimens.

OUTLINE: This is a dose escalation study. Patients receive oral fenretinide once daily on days 1, 8 and 9 and three times a day on days 2-7. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Treatment continues for up to 6 months following complete remission. Accessible tumors are biopsied on day 8. Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 21 patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid malignant tumors (carcinoma or sarcoma) Not eligible for any known treatment or regimen of higher potential efficacy No history of CNS tumors or prior CNS metastases

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/mL SGOT/SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/mL OR Creatinine clearance at least 60 mL/min Cardiovascular: At least 6 months since any acute myocardial infarction No congestive heart failure No New York Heart Association class III or IV heart disease No clinically significant cardiac arrhythmias Pulmonary: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No gastrointestinal bleeding or bleeding tendency

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (at least 6 weeks since nitrosoureas or mitomycin) and recovered No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: No prior systemic retinoid therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1998-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and toxicities of 4-HPR | per cycle
  When drug is administered orally three times daily for 21 doses, repeated every 21 days.

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of 4-HPR and its metabolite(s) | Pre-treatment; Cycle 1 Days 1 & 8: 1, 2, 4, 6, 8, 12, 24 hrs & day

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. LoRusso, DO, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States